CLINICAL TRIAL: NCT00004359
Title: Phase II Pilot Study of Extracorporeal Phototherapy for Epidermolysis Bullosa Acquisita
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Northwestern University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11928; NU-511
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-01

CONDITIONS: Epidermolysis Bullosa Acquisita
Keywords: dermatologic disorders; epidermolysis bullosa; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — Epidermolysis Bullosa Acquisita; Skin Diseases; Epidermolysis Bullosa; Genetic Diseases, Inborn; Rare Diseases | interventions — Methoxsalen

INTERVENTIONS:
Drug: methoxsalen

SUMMARY:
OBJECTIVES: I. Evaluate immunomodulation with extracorporeal photochemotherapy (ECP) in patients with epidermolysis bullosa acquisita.

II. Investigate the effect of ECP on lymphocyte activity.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Oral methoxsalen (8-MOP) is administered 90 minutes prior to leukapheresis. Blood mononuclear cells are exposed to ultraviolet A light for 3 hours, then returned to the patient. The process is repeated on 2 successive days.

Patients are re-treated every 3 to 4 weeks for a total of 6 treatments or until the skin has cleared.

ELIGIBILITY:
* Active epidermolysis bullosa acquisita

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 1996-02

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth B. Gordon, Study Chair — Northwestern University